CLINICAL TRIAL: NCT05314426
Title: Mayo Clinic Phage Program Biobank
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gina A. Suh, Principal Investigator, Mayo Clinic
Other Study IDs: 21-013112
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Bacteriophage Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — whole blood and synovial fluid will be stored in the biorepository for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to help scientists and clinicians discover answers to research questions related to antibiotic-resistant bacterial infections, and the role that phage therapy plays as a possible treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Able to provide informed consent.
* Individual must have a future treatment plan to receive or has historically received phage therapy.

Exclusion Criteria:

* Individuals , 18 years of age.
* Unwilling/unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic patients receiving bacteriophage therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Enrollment of study participants | 5 years
  To recruit and enroll participants up to 100 participants who have received or will receive phage therapy treatment
Collection of biospecimens | 5 years
  Total number of biospecimens collected which may include blood samples and synovial fluid
Medical record review | 5 years
  Review the medical record of enrolled participants to ascertain any new health outcomes.
Increase treatment options and level of care for patients with bacterial infections | 5 years
  Total number of collaborations with clinical investigators and researchers at both Mayo Clinic and across the globe.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Suh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials